CLINICAL TRIAL: NCT04173156
Title: Treatment of Localized Advanced Periodontitis Using an Oscillating Chitosan Device Versus Regular Curettes Alone - a Randomized Parallel Arm Clinical Trial
Brief Title: Treatment of Advanced Periodontitis Using an Oscillating Chitosan Device Versus Regular Curettes Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Labrida AS (Industry)
Responsible Party: Principal Investigator, Caspar Wohlfahrt, Specialist in periodontology, Labrida AS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 256756:2
Record Dates: First submitted 2018-08-16; First posted 2019-11-21 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Examiners blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oscillating Chitosan Device (Experimental): The brush bristles of the test device (Labrida BioClean®, LABRIDA AS, Oslo, Norway) are made of the biopolymer chitosan. Any debris left from the chitosan bristles is completely biocompatible and will dissolve or be resorbed, thus not causing harm to the tissues.surrounding the tooth. Chitosan is made from chitin derived from shell of marine crustaceans such as shrimp and crab, however chemically modified and thus not even considered to be animally derived. Chitosan has been approved for use in e.g., surgical bandages, as a haemostatic agent and as dietary supplement used in a wide range of nutritional and health products. Chitosan has also been documented to be non-allergenic and it has been suggested that chitosan has anti-inflammatory properties.
  Interventions: Device: Labrida Bioclean
- Regular Curettes (Active Comparator): Standard non surgical treatment of active periodontal disease includes supra and subgingival scaling and root planing with periodontal medical grade Gracey system steel curettes
  Interventions: Device: Gracey Periodontal curettes

INTERVENTIONS:
Device: Labrida Bioclean — The brush bristles of the test device (Labrida BioClean®, LABRIDA, Oslo, Norway) are made of the biopolymer chitosan
  Other Names: Gracey Periodontal curettes
  Arms: Oscillating Chitosan Device
Device: Gracey Periodontal curettes — Regular commercially available area specific and medical grade steel Gracey periodontal curettes
  Arms: Regular Curettes

SUMMARY:
40 patients diagnosed with localised periodontitis will be included at each center, 20 patients will be treated with the control treatment, 20 patients will be treated by test treatment.

DETAILED DESCRIPTION:
2.3 This will be a prospective multicentre parallel arm randomized clinical trial of 6 months' duration. Clinical parameters of periodontal disease will be recorded at baseline and at 6 months. Radiographs will be taken at baseline and at 6 months.Treatment will be performed at baseline and thereafter every three months.

2.5 Study setting Patient screening, inclusions and all clinical examinations will be performed by a board-certified specialist in periodontology at the test centres. Treatment will be performed by a registered separate therapist, either dentist or dental hygienist.

2.7 Treatment allocation Patients will be allocated to one of the following treatments: control (curettes+ ultrasound scaler (USS) supra and subgingivally), test (curettes + USS supra and chitosan brush in oscillating handpiece subgingivally) by computer-generated block randomization to ensure equal sample sizes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Periodontitis as previously defined on at least three teeth but less than 8 teeth.

  2. Above 18 years of age.

  3. Eligible for treatment in an outpatient dental clinic (ie, American Society of Anesthesiologist index (ASA) I and II).

  4. Had full-mouth plaque scores ≤ 20% prior to final inclusion3 5. Signed Informed Consent obtained prior to start.

  6. Psychological appropriateness 7. Consent to complete all follow-up visits

Exclusion Criteria:

1. Prosthetic constructions with technical complications which according to the examiners judgement has contributed to the disease state and not possible to resolve prior to final inclusion.
2. Receiving systemic antibiotics < 3 months prior to study start.
3. Pregnant or lactating.
4. Any condition or current treatment for any condition, which in the opinion of the investigator and/or consulting physician, may constitute an unwarranted risk.
5. Presence of psychological characteristics such as inappropriate attitude or motivation which, in the opinion of the investigator, are incompatible with the protocol.
6. Unwillingness to undergo treatment.
7. Ongoing or previous radiotherapy to the head-neck region.
8. Ongoing chemotherapy.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Difference between groups in clinical signs of inflammation | 6 months
  Difference between test and control groups in change in inflammation tested by measuring pocket probing depth (PPD) and Bleeding on Probing (BoP). Probing pocket depths will be recorded at 6 sites around each included tooth using a regular mm scale periodontal probe according to the examiners preferences. Bleeding on probing at the included sites will be assessed using a three-graded index within 30 seconds following probing of the pocket. A score of 0 represented no bleeding, 1 represented isolated minimal bleeding spots, 2 represented blood forming a confluent red line on the margin and 3 represented heavy or profuse bleeding This will be done to assess the clinical efficacy of the Labrida BioClean® biodegradable brush used as mechanical debridement device for treatment of advanced periodontal disease (2017 World Workshop Stage III and IV Grade B). Primary end-point is reduction in periodontal disease as measured clinically up to three months after therapy.

SECONDARY OUTCOMES:
Difference between groups in clinical and radiographic attachment loss | 6 months
  Difference between test and control groups in change in periodontal attachment loss tested by measuring clinical attachment loss and bone level differences on radiographs. This will be done to assess safety of Labrida BioClean® by evaluating the occurrence of adverse events. attachment level (CAL) measurements and radiographs. CAL will be assessed using a regular periodontal mm graded probe (Michigan O with Williams marking) with a force of approximately 20 N (experienced periodontal examiner). Bone attachement on intraoral radiographs at baseline and 6 and 12 months will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Caspar Wohlfahrt, Study Director — Bjerke Tannmedisin
Locations (3):
- Norway (2):
  - Bjerke tannmedisin, Oslo
  - Colosseum Sola, Stavanger
- Yeditetepe University; School of dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No